CLINICAL TRIAL: NCT01778569
Title: Human Translational Studies of Inflammation and Cardiometabolic Diseases: The Psoriasis, Atherosclerosis and Cardiometabolic Disease (PACI) Initiative
Brief Title: The Psoriasis, Atherosclerosis, and Cardiometabolic Disease Initiative (PACI)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130065; 13-H-0065
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-03-20

CONDITIONS: Metabolic Disease; Cardiovascular Disease; Inflammation; Psoriasis
Keywords: Imaging; Cardiovascular Risk Factors; Inflammation; Lipoproteins; Metabolic Dysfunction; Natural History
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases; Inflammation; Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patient with a diagnosis of chronic plaque psoriasis, psoriatic arthritis, or pustular psoriasis

SUMMARY:
Background:

- Cardiometabolic diseases are medical disorders that can occur together and affect the heart. They increase the risk of developing heart disease and diabetes. One disorder, psoriasis, is an inflammation that mostly affects the skin but can affect the entire body. Another disorder, atherosclerosis, is a process in which cholesterol is gradually deposited on the wall of arteries. This causes arteries to harden and become less flexible. Many cells that cause psoriasis also cause atherosclerosis. Researchers want to look at the relationship between cardiometabolic diseases and psoriasis.

Objectives:

- To study the relationship between psoriasis and cardiometabolic diseases.

Eligibility:

- Individuals at least 18 years of age who have psoriasis.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have up to seven outpatient visits over the 4 years. The first visit will be a screening visit. Visits 2 will be12 months after visit 1. Visits 3, 4, and 5, will be scheduled yearly for the next 3 years. If participants have a psoriasis flare with more severe symptoms, they may have an extra visit. Those who leave the study early will have a final visit with the full series of tests.
* At visits 1, 2,and 5, and any flare visits, participants will have a physical exam and medical history. They will provide blood and urine samples, as well as optional tissue biopsies. They will also have heart function tests. Imaging studies, as well as optional photographs of affected areas, will be performed. These tests will also be performed at the final visit.
* At visits 3 and 4, participants will have a physical exam and medical history. They will also provide blood and urine samples, and have heart function tests.

DETAILED DESCRIPTION:
Over the past two decades, inflammation has been identified as an important pathogenic process in cardiometabolic diseases (CMD) such atherosclerotic cardiovascular disease (CVD), dyslipidemia, insulin resistance, diabetes and obesity. However, mechanistic links between inflammation and these disease states in humans remain poorly understood. In this study, we propose to utilize psoriasis, a common, chronic inflammatory T-cell skin disease associated with increased CVD and CMD as a model to understand the effect of chronic inflammation on these diseases states. We will conduct a prospective cohort study to understand the effect of chronic inflammation on vascular and metabolic disease at the NIH Clinical Center. Furthermore, we will initiate a large scale collection of blood and skin from extramural sites to facilitate discovery of pathways involved in inflammatory modulation of CVD and CMD.

ELIGIBILITY:
* INCLUSION CRITERIA
* 18 years of age or older
* Diagnosed with psoriasis clinically confirmed by provider, consisting of typical skin findings and associated findings of systemic disease of joints, nails and hair)

EXCLUSION CRITERIA

* For skin and adipose biopsy, any subject with known bleeding disorder, current fever or on anticoagulation.
* Pregnant women and lactating women, may not undergo any study procedures until they are no longer pregnant or breast feeding.
* Subjects with a contraindication to MRI scanning will not receive the optional PET/MRI. These contraindications include subjects with the following devices:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker or defibrillator
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump
  * Metal shrapnel or bullet
* Subjects with a BMI >45 will also not receive the PET MRI.
* Subjects with severe renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m^2 body surface area according to the Modification of Diet in Renal Disease criteria, will not receive the cardiac CT angiography, or gadolinium contrast agent during the PET/MRI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with a diagnosis of chronic plaque psoriasis, psoriatic arthritis, or pustular psoriasis will be considered for this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Our primary outcome of interest is vascular inflammation measured by standard uptake values from PET-CT imaging with FDG. | 4-6 years
  vascular inflammation measured by standard uptake values from PET-CT imaging with FDG.

SECONDARY OUTCOMES:
Mean Aortic Wall Thickness | 4-6 years
Coronary Artery Calcium Score | 4-6 years
HDL function | 4-6 years
lipoprotein particle size and number | 4-6 years
immune, metabolic & inflammation measure | 4-6 years
Myocardial Flow Reserve (MFR) | 4-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Florida EM, Li H, Hong CG, Ongstad EL, Gaddipati R, Sitaula S, Varma V, Parel PM, O'Hagan R, Chen MY, Teague HL, Playford MP, Karathanasis SK, Collen A, Mehta NN, Remaley AT, Sorokin AV. Relationship of Soluble Lectin-Like Low-Density Lipoprotein Receptor-1 (sLOX-1) With Inflammation and Coronary Plaque Progression in Psoriasis. J Am Heart Assoc. 2023 Nov 21;12(22):e031227. doi: 10.1161/JAHA.123.031227. Epub 2023 Nov 20. PMID 37982276
- [Derived] Sorokin AV, Patel N, Li H, Hong CG, Sampson M, O'Hagan R, Florida EM, Teague HL, Playford MP, Chen MY, Mehta NN, Remaley AT. Estimated sdLDL-C for predicting high-risk coronary plaque features in psoriasis: a prospective observational study. Lipids Health Dis. 2023 Apr 27;22(1):55. doi: 10.1186/s12944-023-01819-x. PMID 37106374
- [Derived] Teague HL, Li H, Berg AR, Hong C, Petrole RF, O'Hagan R, Florida EM, Keel A, Rodante J, Kapoor P, Gonzalez-Cantero A, Sorokin AV, Joshi A, Patel N, Gelfand JM, Playford MP, Mehta NN. The Relationship between Circulating APOA-1 and Atherosclerosis Initiation and Progression in Psoriasis. J Invest Dermatol. 2023 Oct;143(10):1947-1954.e4. doi: 10.1016/j.jid.2023.01.044. Epub 2023 Apr 22. PMID 37088280
- [Derived] Sajja A, Abdelrahman KM, Reddy AS, Dey AK, Uceda DE, Lateef SS, Sorokin AV, Teague HL, Chung J, Rivers J, Joshi AA, Elnabawi YA, Goyal A, Rodante JA, Keel A, Alvarez JE, Lockshin B, Prussick R, Siegel E, Playford MP, Chen MY, Bluemke DA, Gelfand JM, Mehta NN. Chronic inflammation in psoriasis promotes visceral adiposity associated with noncalcified coronary burden over time. JCI Insight. 2020 Nov 19;5(22):e142534. doi: 10.1172/jci.insight.142534. PMID 33104056
- [Derived] Salahuddin T, Natarajan B, Playford MP, Joshi AA, Teague H, Masmoudi Y, Selwaness M, Chen MY, Bluemke DA, Mehta NN. Cholesterol efflux capacity in humans with psoriasis is inversely related to non-calcified burden of coronary atherosclerosis. Eur Heart J. 2015 Oct 14;36(39):2662-5. doi: 10.1093/eurheartj/ehv339. Epub 2015 Jul 18. PMID 26188212
- [Derived] Rose S, Stansky E, Dagur PK, Samsel L, Weiner E, Jahanshad A, Doveikis J, Naik HB, Playford MP, McCoy JP, Mehta NN. Characterization of immune cells in psoriatic adipose tissue. J Transl Med. 2014 Sep 16;12:258. doi: 10.1186/s12967-014-0258-2. PMID 25224267
- [Derived] Mehta NN, Dagur PK, Rose SM, Naik HB, Stansky E, Doveikis J, Biancotto A, Playford MP, Philip McCoy J Jr. IL-17A production in human psoriatic blood and lesions by CD146+ T cells. J Invest Dermatol. 2015 Jan;135(1):311-314. doi: 10.1038/jid.2014.317. Epub 2014 Jul 24. No abstract available. PMID 25058615
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-H-0065.html